CLINICAL TRIAL: NCT03749096
Title: IVIg in Glycine Receptor Antibody Positive Stiff-person Syndrome (SPS) Spectrum Disorders.
Brief Title: Randomized Placebo Controlled Trial of IVIg in Glycine Receptor Antibody Positive Stiff-person Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment did not meet sponsors timeline
Sponsor: Mayo Clinic (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Andrew McKeon, Prinicple Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-007041
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Stiff-Person Syndrome
Keywords: IVIG; stiff-person syndrome; SPS; glycine receptor antibody; intravenous immunoglobulin; GlyRα1
MeSH Terms: conditions — Stiff-Person Syndrome | interventions — Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous immunoglobulin (Active Comparator): IVIg dose will be 2g/kg ideal body weight every 4 weeks (in 2 divided doses on consecutive days) for 12 weeks (3 cycles total).
  Interventions: Drug: Intravenous Immunoglobulins, Human
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Intravenous Immunoglobulins, Human — Immunoglobulins are fractionated blood products made from pooled human plasma.
  Arms: Intravenous immunoglobulin
Drug: Placebos — Normal Saline
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This is a randomized double-blind controlled trial of intravenous immunoglobulin (IVIg) for glycine receptor antibody positive (GlyRα1) antibody Stiff Person Syndrome (SPS) spectrum disorders. Adult patients will be enrolled over the course of 36 months. Study duration per patient will be 11 weeks. Total study duration will be 39 months. All treatment and study visits will occur at Mayo Clinic in Rochester, MN.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether intravenous immunoglobulin (IVIG) treatment reduces stiffness and spasms in patients with SPS spectrum disorders compared to patients who do not receive any treatment. In this study, investigators want to compare the effects, good and/or bad, of IVIG with placebo on participants with SPS to find out which is better. This is a "randomized, double-blind" study. Which treatment participants will receive is randomly determined. Participants have an equal chance of receiving IVIG or the placebo.

SPS spectrum cohort will include any from the SPS spectrum patient (stiff-limbs, stiff-trunk, stiff-limbs and trunk, and PERM). Study visits will be considered part of clinical care and will occur at: enrollment (will coincide with screening visit), and 11 weeks. IVIg/placebo (saline) treatments will be administered on 2 consecutive days in week 1, week 5, week 9 in all patients.

ELIGIBILITY:
Inclusion Criteria

* Patient must be 18 years of age or older
* Must have symptoms of SPS for less than 3 years
* If taking corticosteroids, the patients must be on a stabile dose for 30 days prior to enrolment
* Patients will have a diagnosis of SPS spectrum disorder based on both of clinical and serological status

Exclusion Criteria

* Patients on immune suppressants initiated/dose increased in the prior 6 months
* History of thrombotic episodes within the 2 years prior to enrollment
* Known allergic or other severe reactions to blood products including intolerability to previous IVIG
* Previous adequate trial of IVIG as determined by the Principal Investigator
* IgA deficiency
* Reproductive status:

  * Women who are pregnant, breastfeeding
  * Women and men of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period, as evaluated by the investigator.
* Any surgical procedure within 4 weeks prior to baseline.
* Evidence of serious uncontrolled concomitant diseases that may preclude patient participation; Other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency
* Known active infection within 4 weeks prior to baseline.
* Evidence of chronic active hepatitis B or C.
* Active ischemic heart disease in the past year prior to baseline.
* Patients should not have severe renal or hepatic disease
* Severe hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Distribution-of-stiffness index | Screen, Week 11
  Scores on this index range from 0 to 6 and reflect the extent of stiffness. with One point being given for stiffness in each of the following areas: lower trunk, upper trunk, legs, arms, face, and abdomen. Lower scores indicate less stiffness.
Change in Heightened-sensitivity scale | Screen, Week 11
  Scores range from 1 to 7 based on response; one point being given for each source of or type of spasm, as follows: unexpected noises, visual stimuli, somatosensory stimuli, voluntary activities, emotional upset or stress, no specific stimuli, and nocturnal spasms. Lower scores indicate less frequent spasms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McKeon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States